CLINICAL TRIAL: NCT00056836
Title: A Phase III, Multicenter, Randomized, Double Masked, Sham Injection-Controlled Study of the Efficacy and Safety of rhuFab V2 (Ranibizumab) in Subjects With Minimally Classic or Occult Subfoveal Neovascular Age-Related Macular Degeneration
Brief Title: A Study to Evaluate rhuFab V2 in Subjects With Minimally Classic or Occult Subfoveal Neovascular Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: FVF2598g
Record Dates: First submitted 2003-03-24; First posted 2003-03-26 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Macular Degeneration
Keywords: AMD; Neovascular age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

INTERVENTIONS:
Drug: rhuFab V2 (ranibizumab)

SUMMARY:
The purpose of this study is to determine whether injections of rhuFab V2 into the eye can prevent vision loss in patients with age-related macular degeneration, and also to evaluate the safety of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age >=50 years
* Active primary or recurrent subfoveal choroidal neovascularization (CNV) lesions secondary to age-related macular degeneration (AMD) in the study eye
* Lesions with occult CNV or with some classic CNV component are permissible. However, if classic CNV (well-demarcated hyperfluorescence boundaries in the early phase of the fluorescein angiogram) is present, the area of classic CNV must be <50% of the total lesion size.
* The total area of CNV (including both classic and occult components) encompassed within the lesion must be >=50% of the total lesion area.
* The total lesion area must be <=12 disc areas (DA) in size.
* Best corrected visual acuity, using Early Treatment of Diabetic Retinopathy Study (ETDRS) charts, of 20/40 to 20/320 (Snellen equivalent) in the study eye

Exclusion Criteria:

* Prior treatment with verteporfin, external-beam radiation therapy, or transpupillary thermotherapy (TTT) in the study eye
* Treatment with verteporfin in the non-study eye less than 7 days preceding Day 0
* Previous participation in a clinical trial (for either eye) involving anti-angiogenic drugs (pegaptanib, ranibizumab, anecortave acetate, protein kinase C inhibitors, etc.)
* Previous intravitreal drug delivery (e.g., intravitreal corticosteroid injection or device implantation) in the study eye
* Previous subfoveal focal laser photocoagulation in the study eye
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1 month preceding Day 0
* History of vitrectomy surgery in the study eye
* History of submacular surgery or other surgical intervention for AMD in the study eye
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals)
* Subretinal hemorrhage in the study eye that involves the center of the fovea, if the size of the hemorrhage is either >=50% of the total lesion area or >=1 disc area in size
* Subfoveal fibrosis or atrophy in the study eye
* CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia
* Retinal pigment epithelial tear involving the macula in the study eye
* Any concurrent intraocular condition in the study eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, could either: (1) Require medical or surgical intervention during the 24-month study period to prevent or treat visual loss that might result from that condition, or (2) If allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of best corrected visual acuity over the 24-month study period
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia or absence of the posterior capsule in the study eye
* Spherical equivalent of the refractive error in the study eye demonstrating more than -8 diopters of myopia
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding Day 0
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure >= 30 mmHg despite treatment with anti-glaucoma medication)
* History of glaucoma filtering surgery in the study eye
* History of corneal transplant in the study eye
* Premenopausal women not using adequate contraception
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications
* Current treatment for active systemic infection
* History of allergy to fluorescein, not amenable to treatment
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed and graded by the central reading center
* Inability to comply with study or follow up procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720
Dates: Start 2003-03; Study Completion 2005-12 (Actual)

REFERENCES:
- [Result] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Result] Suner IJ, Kokame GT, Yu E, Ward J, Dolan C, Bressler NM. Responsiveness of NEI VFQ-25 to changes in visual acuity in neovascular AMD: validation studies from two phase 3 clinical trials. Invest Ophthalmol Vis Sci. 2009 Aug;50(8):3629-35. doi: 10.1167/iovs.08-3225. Epub 2009 Feb 28. PMID 19255158
- [Derived] Blodi BA, Domalpally A, Corkery E, Osborne A, Blotner S, Grzeschik SM, Gune S. Prevalence of Macular Atrophy in the MARINA Study of Ranibizumab versus Sham for Neovascular Age-Related Macular Degeneration. Ophthalmol Retina. 2023 Aug;7(8):661-671. doi: 10.1016/j.oret.2023.03.004. Epub 2023 Apr 22. PMID 37086257
- [Derived] Mollan SP, Fu DJ, Chuo CY, Gannon JG, Lee WH, Hopkins JJ, Hughes C, Denniston AK, Keane PA, Cantrell R. Predicting the immediate impact of national lockdown on neovascular age-related macular degeneration and associated visual morbidity: an INSIGHT Health Data Research Hub for Eye Health report. Br J Ophthalmol. 2023 Feb;107(2):267-274. doi: 10.1136/bjophthalmol-2021-319383. Epub 2021 Sep 13. PMID 34518162
- [Derived] Weinberg DV, Shapiro H, Ehrlich JS. Ranibizumab treatment outcomes in phakic versus pseudophakic eyes: an individual patient data analysis of 2 phase 3 trials. Ophthalmology. 2013 Jun;120(6):1278-82. doi: 10.1016/j.ophtha.2012.11.042. Epub 2013 Feb 28. PMID 23453513
- [Derived] Xu L, Lu T, Tuomi L, Jumbe N, Lu J, Eppler S, Kuebler P, Damico-Beyer LA, Joshi A. Pharmacokinetics of ranibizumab in patients with neovascular age-related macular degeneration: a population approach. Invest Ophthalmol Vis Sci. 2013 Mar 5;54(3):1616-24. doi: 10.1167/iovs.12-10260. PMID 23361508
- [Derived] Bressler NM, Chang TS, Varma R, Suner I, Lee P, Dolan CM, Ward J, Ianchulev T, Fine J. Driving ability reported by neovascular age-related macular degeneration patients after treatment with ranibizumab. Ophthalmology. 2013 Jan;120(1):160-8. doi: 10.1016/j.ophtha.2012.07.027. Epub 2012 Sep 23. PMID 23009891
- [Derived] Elshout M, van der Reis MI, Webers CA, La Heij EC, Hendrikse F, Schouten JS. A new epidemiological aid in deciding whether to continue or stop a treatment. Invest Ophthalmol Vis Sci. 2012 Jul 1;53(8):4331-6. doi: 10.1167/iovs.11-9242. PMID 22661474
- [Derived] Rosenfeld PJ, Shapiro H, Ehrlich JS, Wong P; MARINA and ANCHOR Study Groups. Cataract surgery in ranibizumab-treated patients with neovascular age-related macular degeneration from the phase 3 ANCHOR and MARINA trials. Am J Ophthalmol. 2011 Nov;152(5):793-8. doi: 10.1016/j.ajo.2011.04.025. Epub 2011 Jul 26. PMID 21794843
- [Derived] Hawkins BS, Bressler NM, Reynolds SM. Patient-reported outcomes among sham vs no-treatment controls from randomized trials. Arch Ophthalmol. 2011 Feb;129(2):200-5. doi: 10.1001/archophthalmol.2010.359. PMID 21320967
- [Derived] Rosenfeld PJ, Shapiro H, Tuomi L, Webster M, Elledge J, Blodi B; MARINA and ANCHOR Study Groups. Characteristics of patients losing vision after 2 years of monthly dosing in the phase III ranibizumab clinical trials. Ophthalmology. 2011 Mar;118(3):523-30. doi: 10.1016/j.ophtha.2010.07.011. PMID 20920825
- [Derived] Barbazetto I, Saroj N, Shapiro H, Wong P, Freund KB. Dosing regimen and the frequency of macular hemorrhages in neovascular age-related macular degeneration treated with ranibizumab. Retina. 2010 Oct;30(9):1376-85. doi: 10.1097/IAE.0b013e3181dcfb0b. PMID 20683380
- [Derived] Barbazetto IA, Saroj N, Shapiro H, Wong P, Ho AC, Freund KB. Incidence of new choroidal neovascularization in fellow eyes of patients treated in the MARINA and ANCHOR trials. Am J Ophthalmol. 2010 Jun;149(6):939-946.e1. doi: 10.1016/j.ajo.2010.01.007. Epub 2010 Apr 8. PMID 20378094
- [Derived] Bressler NM, Chang TS, Suner IJ, Fine JT, Dolan CM, Ward J, Ianchulev T; MARINA and ANCHOR Research Groups. Vision-related function after ranibizumab treatment by better- or worse-seeing eye: clinical trial results from MARINA and ANCHOR. Ophthalmology. 2010 Apr;117(4):747-56.e4. doi: 10.1016/j.ophtha.2009.09.002. Epub 2010 Mar 2. PMID 20189654
- [Derived] Chang TS, Bressler NM, Fine JT, Dolan CM, Ward J, Klesert TR; MARINA Study Group. Improved vision-related function after ranibizumab treatment of neovascular age-related macular degeneration: results of a randomized clinical trial. Arch Ophthalmol. 2007 Nov;125(11):1460-9. doi: 10.1001/archopht.125.11.1460. PMID 17998507